CLINICAL TRIAL: NCT05318118
Title: Comparative of Clinical and Evaluation Results of Medial Meniscus Arthroscopic Reconstruction Using the Fast Fix and FiberStitch Systems
Brief Title: Comparison of the Results of Arthroscopic Suturing of the Medial Meniscus Using the Fast Fix and FiberStitch Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: eMKa MED Medical Center (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB-98/2021
Record Dates: First submitted 2021-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Meniscus; Detachment, Current Injury; Detachment; Medial Mensical Tear; Medial Meniscus Knee Injury
Keywords: meniscus;; medial;; injury;; suture;; techniques;
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The results refering to the operated limb will be compared in both groups between themselves and furthermore with the results of clinical and biomechanical studies on non-operated limbs.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial Meniscus Arthroscopic Reconstruction Using the Fast Fix (Active Comparator)
  Interventions: Procedure: Medial Meniscus Arthroscopic Reconstruction Using the Fast Fix
- Medial Meniscus Arthroscopic Reconstruction Using the Fiber Stitch (Active Comparator)
  Interventions: Procedure: Medial Meniscus Arthroscopic Reconstruction Using the Fiber Stitch

INTERVENTIONS:
Procedure: Medial Meniscus Arthroscopic Reconstruction Using the Fast Fix — Arthroscopic reconstruction of damaged Medial Meniscus using Fast-Fix (Smith & Nephew) implant.
  Arms: Medial Meniscus Arthroscopic Reconstruction Using the Fast Fix
Procedure: Medial Meniscus Arthroscopic Reconstruction Using the Fiber Stitch — Arthroscopic reconstruction of damaged Medial Meniscus using Fiber-Stitch (Arthrex) implant
  Arms: Medial Meniscus Arthroscopic Reconstruction Using the Fiber Stitch

SUMMARY:
Clinical and comparative evaluation of the treatment results of arthroscopic reconstruction of the medial meniscus of the knee joint using the Fast Fix and FiberStitch systems.

DETAILED DESCRIPTION:
The main goal of the project is to evaluate the results of medial meniscus traumatic injury suturing. Further (detailed) objectives are: to compare the results obtained in the study groups of suturing the medial meniscus with the use of two systems: Fast Fix (smith & nephew) and Fiber Stitch (arthrex). The results refering to the operated limb will be compared in both groups between themselves and furthermore with the results of clinical and biomechanical studies on non-operated limbs.

ELIGIBILITY:
Inclusion Criteria:

* Isolated MM damage.
* Operation performed only in arthroscopy technique.
* No any knee intervention earlier.
* No other pathology in the anatomical area.
* Patient informed consent to participate in research

Exclusion Criteria:

* Age under 18 years old or above 35 years old.
* Any knee intervention performed earlier.
* Any other pathology in the anatomical area identified during preoperative diagnostics.
* Any damage in the area of the second knee joint.
* Failure complying the same treatment protocol rigor.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Tegner Activity Level Scale (TAS); | 1 day
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS); | 3 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS); | 6 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS); | 12 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Visual Analogue Score (VAS) | 1 day
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 3 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 6 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 12 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 1 day
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 3 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 6 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 12 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
Knee Society Score (KSS); | 1 day
  The Knee Society Score (KSS) evaluates the clinical picture in terms of pain intensity, range of motion and stability in the anteroposterior and mediolateral planes, flexion deformities, contractures and poor alignment, and is widely used in clinic and mentioned in orthopedic literature.
  Grading for the Knee Society Score:
  * 80-100 - excellent;
  * 70-79 - good;
  * 60-60 - fair;
  * below 60 - poor.
Knee Society Score (KSS); | 3 months after procedure
  The Knee Society Score (KSS) evaluates the clinical picture in terms of pain intensity, range of motion and stability in the anteroposterior and mediolateral planes, flexion deformities, contractures and poor alignment, and is widely used in clinic and mentioned in orthopedic literature.
  Grading for the Knee Society Score:
  * 80-100 - excellent;
  * 70-79 - good;
  * 60-60 - fair;
  * below 60 - poor.
Knee Society Score (KSS); | 6 months after procedure
  The Knee Society Score (KSS) evaluates the clinical picture in terms of pain intensity, range of motion and stability in the anteroposterior and mediolateral planes, flexion deformities, contractures and poor alignment, and is widely used in clinic and mentioned in orthopedic literature.
  Grading for the Knee Society Score:
  * 80-100 - excellent;
  * 70-79 - good;
  * 60-60 - fair;
  * below 60 - poor.
Knee Society Score (KSS); | 12 months after procedure
  The Knee Society Score (KSS) evaluates the clinical picture in terms of pain intensity, range of motion and stability in the anteroposterior and mediolateral planes, flexion deformities, contractures and poor alignment, and is widely used in clinic and mentioned in orthopedic literature.
  Grading for the Knee Society Score:
  * 80-100 - excellent;
  * 70-79 - good;
  * 60-60 - fair;
  * below 60 - poor.
Knee Injury and Osteoarthritis Outcome Score (KOOS); | 1 day
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee.
  It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Knee Injury and Osteoarthritis Outcome Score (KOOS); | 3 months after procedure
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee.
  It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Knee Injury and Osteoarthritis Outcome Score (KOOS); | 6 months after procedure
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee.
  It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Knee Injury and Osteoarthritis Outcome Score (KOOS); | 12 months after procedure
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee.
  It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Tegner Lysholm Knee Scoring Scale; | 1 day
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale; | 3 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale; | 6 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale; | 12 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Body Mass Index (BMI) | 1 day
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 3 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 6 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 12 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Biomechanical examination | 9 months after procedure
  On the Biodex 3 System measuring device
Biomechanical examination | 12 months after procedure
  On the Biodex 3 System measuring device
Ultrasound examination (USG) | 6 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry
Ultrasound examination (USG) | 12 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry
Magnetic resonance imaging (MRI) | 6 months after procedure
  1,5 Tesli
Magnetic resonance imaging (MRI) | 12 months after procedure
  1,5 Tesli

CONTACTS AND LOCATIONS:
Locations (1):
- eMKa MED Medical Center, Wroclaw, Dolnośląsk, Poland

IPD SHARING:
Plan to Share IPD: No